CLINICAL TRIAL: NCT06771011
Title: Prospective Comparative Validation Study of RUCAM and RECAM
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MR-11-23-024371
Record Dates: First submitted 2024-08-22; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Drug Induced Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A total of 407 hospitalized patients with acute liver injury in Beijing Friendship Hospital Affiliated to Capital Medical University were enrolled. The clinical information, biochemical examination, imageological examination (ultrasound, CT, MRI) and liver biopsy pathology of patients with acute liver injury will be collected. The diagnostic efficacy of RECAM and RUCAM in the diagnosis of DILI will be compared, and the consistency of different clinicians in the diagnosis of DILI using RECAM and RUCAM scores will also be compared.

DETAILED DESCRIPTION:
Patients admitted to Beijing Friendship Hospital affiliated with Capital Medical University from March 2023 to September 2024 who meet the inclusion criteria will be included in the study. Data collected will include demographic information, clinical manifestations, laboratory tests, imaging examinations, and liver pathology reports. Three clinical doctors will independently score the patients, calculating the RECAM and RUCAM scores to compare the diagnostic efficacy of RECAM and RUCAM, as well as the consistency of the two scoring systems in diagnosing DILI. Additionally, statistical analysis will be performed on patients' clinical manifestations, laboratory tests, imaging examinations, and liver pathology reports.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old
2. Acute liver injury within 3 months of onset and biochemical meeting one of the following criteria: ALT≥5 ULN; ALP≥2 ULN; ALT≥3 ULN and TBil≥2 ULN
3. The patients had a clear history of medication: the time from medication to onset, the time from drug withdrawal to onset, the time of the first laboratory test and the peak laboratory test, the reason for taking medication, the name of the drug, the dose of the drug, and the frequency. If the causative drug includes traditional Chinese medicine, the specific name of all the components or patent Chinese medicine in the prescription, a single drug or single component, or the main ingredient in the prescription causing liver injury should be provided
4. All the key data for RUCAM and RECAM can accurately be contained.
5. Follow-up outcomes confirmed that the cause of the acute liver injury was any of the following liver diseases: Drug-induced liver injury, acute viral hepatitis (including acute viral hepatitis A, acute viral hepatitis B or acute exacerbation of chronic hepatitis B, acute viral hepatitis E), alcoholic liver disease, autoimmune hepatitis, biliary calculi, biliary obstruction, hypoxic-ischemic hepatitis, congestive liver disease and other liver diseases

Exclusion Criteria:

1. The incubation period cannot be accurately calculated: the dates of starting medication, stopping medication, and onset of illness cannot be accurately described, resulting in the inability to calculate the incubation period
2. Can not be clear about the pathogenic drug: the pathogenic drug is only described as "traditional Chinese medicine, cold medicine, antipyretic medicine", but cannot be clear about what kind of medicine
3. Missing biochemical data, resulting in inability to assess the time of 50% decrease in liver biochemistry (ALT or ALP, TBIL) from the peak after drug withdrawal
4. The cause of the patient's acute liver injury could not be determined
5. Acetaminophen liver injury
6. Toxic liver disease, such as mushroom poisoning caused liver damage, chemical poisons (such as paint, etc.) liver damage
7. Previous liver transplantation and bone marrow transplantation
8. Pregnancy or lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population who met the above inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 407 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
RECAM is not inferior to RUCAM | July 2025
  Area under the curve (AUC) values for the identification of DILI cases were compared by the Delong method. The AUROC of RUCAM in diagnosing DILI was higher than RECAM. The pattern of liver injury was classified by the R-value based on the first available liver chemistries. Individual scores of the RUCAM and RECAM were calculated with the appropriate algorithms.
RECAM is inferior to RUCAM | July 2025
  Area under the curve (AUC) values for the identification of DILI cases were compared by the Delong method. The AUROC of RUCAM in diagnosing DILI was higher than RECAM. The pattern of liver injury was classified by the R-value based on the first available liver chemistries. Individual scores of the RUCAM and RECAM were calculated with the appropriate algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Xinyan Zhao, Study Chair — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No